CLINICAL TRIAL: NCT05861427
Title: A Phase 2/3, Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel-Group Study With An Active Treatment Extension to Evaluate the Efficacy, Safety, and Tolerability of Oral Atogepant for the Prevention of Migraine in Japanese Subjects With Episodic Migraine
Brief Title: Study of Oral Atogepant Tablets to Assess Change in Disease Activity in Adult Japanese Participants With Episodic Migraine
Acronym: JPN PIVOTAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M22-056
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Migraine
Keywords: Migraine; Episodic Migraine; Atogepant
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Atogepant Dose A (Experimental): Participants will receive atogepant dose A once daily (QD) for 24 weeks.
  Interventions: Drug: Atogepant
- Atogepant Dose B (Experimental): Participants will receive atogepant dose B QD for 24 weeks.
  Interventions: Drug: Atogepant
- Atogepant Dose C (Experimental): Participants will receive atogepant dose C QD for 24 weeks.
  Interventions: Drug: Atogepant
- Placebo (Experimental): Participants will receive placebo QD for 12 weeks. Participants will be re-randomized at week 12 to receive atogepant dose A, dose B or dose C QD for 12 weeks.
  Interventions: Drug: Atogepant; Drug: Placebo for Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: Qulipta
Drug: Placebo for Atogepant — Oral Tablet
  Arms: Placebo

SUMMARY:
A migraine is a moderate to severe headache on one side of the head. A migraine attack is a headache that may be accompanied by throbbing, nausea, vomiting, sensitivity to light and sound, or other symptoms. This study will assess how safe and effective three different doses of atogepant is compared to placebo in adult Japanese participants. Change in migraine symptoms will be assessed.

Atogepant (Qulipta) is an approved drug to treat adults with episodic migraine in the United States. Participants are randomly assigned to one of the 4 treatment groups called Arms to receive atogepant or matching placebo. There is 1 in a 4 chance for the participant to receive placebo. This is double-blinded study which means neither study doctor not the participant will know if the participant received atogepant or placebo. Approximately 520 adult participants with episodic migraine will be enrolled in approximately 50 sites across Japan.

Participants will receive oral atogepant or matching placebo tablets once daily for 12 weeks. At 12 weeks participants assigned to atogepant dose A, dose B or dose C will continue to receive same treatment for 12 additional weeks and participants assigned to placebo will be re-randomized to receive atogepant dose A, dose B or dose C for 12 additional weeks. All participants will be followed for 30 days following last dose of study drug.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The safety and tolerability of the treatment will be checked by medical assessments, blood tests, checking for adverse events and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine (with or without aura).
* Less than 50 years of age at the time of migraine onset.
* History of 4 to 14 migraine days per month in the 3 months prior to screening.
* 4 to 14 migraine days in the baseline period and completed at least 20 out of 28 days at the baseline period per the eDiary.

Exclusion Criteria:

* Difficulty with distinguishing migraine headaches from tension-type or other headaches.
* Clinically significant hematologic, endocrine, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Mean Monthly Migraine Days | Up to 12 Weeks
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed, as per participant eDiary.
Number of Participants Experiencing With Adverse Events (AEs) | Up to approximately 28 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change From Baseline in Mean Monthly Headache Days | Up to Week 12
  A headache day is defined as any calendar day on which headache pain lasting 2 hours or longer occurs unless an acute headache medication was used after the start of the headache, in which case no minimum duration will be specified.
Change From Baseline in Mean Monthly Acute Medication Use Days | Up to Week 12
  An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) for the acute treatment of migraine.
Percentage of Participants Achieving At Least 50% Reduction in the 3-month Average of Monthly Migraine Days | Up to Week 12
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed, as per participant eDiary.
Change From Baseline in Migraine Specific Quality of Life Questionnaire, Version 2.1 (MSQ v2.1) Role Function-Restrictive Domain Score | Up to Week 12
  MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality of life impairments attributed to migraine in the past 4 weeks. It is divided into three domains: Role Function Restrictive, Role Function Preventive, and Emotional Function domain. Participants respond to items using a 6-point scale ranging from "none of the time" to "all of the time." Raw dimension scores are computed as a sum of item responses and rescaled to a 0 to 100 scale, where higher scores indicate better quality of life.
Change From Baseline in Mean Monthly Performance of Daily Activities Domain Score of the Activity Impairment in Migraine - Diary (AIM-D) | Up to Week 12
  The AIM-D is an 11-item daily diary measure that assesses the impact of migraine and is comprised of two domains that evaluate performance of daily activities (7 items) and physical impairment (4 items). Participants are asked to rate the level of difficulty experienced in the past 24 hours with performance of daily activities and physical impairment using a 6 point rating scale ranging from "Not difficult at all" to "I could not do it at all." Scores range from 0-100 scale, with higher scores indicating greater impact of migraine.
Change From Baseline in Mean Monthly Physical Impairment Domain Score of the AIM-D | Up to Week 12
  The AIM-D is an 11-item daily diary measure that assesses the impact of migraine and is comprised of two domains that evaluate performance of daily activities (7 items) and physical impairment (4 items). Participants are asked to rate the level of difficulty experienced in the past 24 hours with performance of daily activities and physical impairment using a 6 point rating scale ranging from "Not difficult at all" to "I could not do it at all." Scores range from 0-100 scale, with higher scores indicating greater impact of migraine.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (48):
- Japan (48):
  - Tokyo Dental College Ichikawa General Hospital /ID# 247436, Ichikawa-shi, Chiba
  - Takanoko Hospital /ID# 245658, Matsuyama, Ehime
  - Fukuiken Saiseikai Hospital /ID# 245662, Fukui-shi, Fukui
  - Jinnouchi Neurosurgical Clinic /ID# 245510, Kasuga-shi, Fukuoka
  - Ikeda Neurosurgical Clinic /ID# 245881, Kasuga-shi, Fukuoka
  - SUBARU Health Insurance Society Ota Memorial Hospital /ID# 247948, Ota-shi, Gunma
  - Hiroshima City Hiroshima Citizens Hospital /ID# 246683, Hiroshima, Hiroshima
  - Higashi Sapporo Neurology And Neurosurgery Clinic /ID# 245667, Sapporo, Hokkaido
  - Nakamura Memorial Hospital /ID# 247379, Sapporo, Hokkaido
  - Konan Medical Center /ID# 245557, Kobe, Hyōgo
  - Nishinomiya Municipal Central Hospital /ID# 246571, Nishinomiya-shi, Hyōgo
  - Yamaguchi Clinic /ID# 246370, Nishinomiya-shi, Hyōgo
  - Mito Kyodo General Hospital /ID# 245487, Mito, Ibaraki
  - Tsukuba Neurosurgery/Headache Clinic /ID# 254665, Tsukuba, Ibaraki
  - Kijima Neurosurgery Clinic /ID# 245758, Kahoku-gun, Ishikawa-ken
  - Kanazawa Neurosurgical Hospital /ID# 254210, Nonoichi-shi, Ishikawa-ken
  - Tokai University Hospital /ID# 245971, Isehara, Kanagawa
  - Fujitsu Clinic /ID# 245811, Kawasaki-shi, Kanagawa
  - Atago Hospital /ID# 245818, Kochi, Kochi
  - Umenotsuji Clinic /ID# 246103, Kochi, Kochi
  - Saiseikai Kumamoto Hospital /Id# 253546, Kumamoto, Kumamoto
  - Narikawa Neurological Clinic /ID# 254023, Sendai, Miyagi
  - Sendai Headache and Neurology Clinic Medical Corporation /ID# 245664, Sendai, Miyagi
  - Makabe Clinic /ID# 246621, Okayama, Okayama-ken
  - Okayama City General Medical Center /ID# 246007, Okayama, Okayama-ken
  - Gokeikai Osaka Kaisei Hospital /ID# 246623, Osaka, Osaka
  - Chibune General Hospital /ID# 245973, Osaka, Osaka
  - Tominaga Clinic /ID# 245812, Osaka, Osaka
  - Takase Internal Medicine Clinic /ID# 245532, Toyonaka-shi, Osaka
  - Saitama Medical University Hospital /ID# 245663, Iruma-gun, Saitama
  - Saino Clinic /ID# 245921, Tokorozawa-shi, Saitama
  - Japanese Red Cross Shizuoka Hospital /ID# 246204, Shizuoka, Shizuoka
  - Dokkyo Medical University Hospital /ID# 246472, Mibu, Tochigi
  - Tokai University Hachioji Hospital /ID# 248326, Hachioji-shi, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 246470, Minato-ku, Tokyo
  - Usuda Clinic Of Internal Medicine /ID# 246166, Setagaya-ku, Tokyo
  - Tokyo Headache Clinic /ID# 245486, Shibuya-ku, Tokyo
  - Keio University Hospital /ID# 245660, Shinjuku-ku, Tokyo
  - Suzuki Kei Yasuragi Clinic /ID# 253493, Tachikawa-shi, Tokyo
  - Sakura neuro Clinic /ID# 248320, Toyama, Toyama
  - Tendo Brain Clinic /ID# 246205, Tendo-shi, Yamagata
  - Nagaseki Headache Clinic /ID# 245485, Kai, Yamanashi
  - DOI Internal Medicine-Neurology Clinic /ID# 245661, Hiroshima
  - Tanaka Neurosurgical Clinic /ID# 245488, Kagoshima
  - Tatsuoka Neurology Clinic /ID# 245328, Kyoto
  - Ooba Clinic for Neurosurgery & Headache /ID# 246201, Ōita
  - Kokubu Clinic /ID# 245810, Takamatsu
  - Shinagawa Strings Clinic /ID# 245665, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Matsumori Y, Yamada H, Nagaseki Y, Shimizu K, Nagy K, Matsuzawa R, Otani T, He MY, Guo H, Ahmadyar G, Takeshima T. Atogepant for the preventive treatment of episodic migraine in Japanese participants: A phase 2/3, randomized, double-blind, placebo-controlled trial with an active treatment extension (RELEASE). Cephalalgia. 2025 Sep;45(9):3331024251374569. doi: 10.1177/03331024251374569. Epub 2025 Sep 26. PMID 41002192
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-056